CLINICAL TRIAL: NCT00004139
Title: Phase II Randomized Trial of Gemcitabine/Docetaxel and Gemcitabine/Irinotecan in Stage IIIB/IV Non-Small Cell Lung Cancer
Brief Title: Gemcitabine Plus Docetaxel or Irinotecan in Treating Patients With Stage IIIB or Stage IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-39809; U10CA031946 (NIH); CLB-39809; CDR0000067369 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 1999-12-10; First posted 2004-05-25 (Estimated); Last update posted 2016-07-20 (Estimated); Status verified 2016-07

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Docetaxel; Gemcitabine; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine + Irinotecan (Experimental)
  Interventions: Drug: gemcitabine hydrochloride; Drug: irinotecan hydrochloride
- Gemcitabine + Docetaxel (Experimental)
  Interventions: Drug: docetaxel; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: docetaxel
  Arms: Gemcitabine + Docetaxel
Drug: gemcitabine hydrochloride
Drug: irinotecan hydrochloride
  Arms: Gemcitabine + Irinotecan

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to compare the effectiveness of gemcitabine plus either docetaxel or irinotecan in treating patients who have stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the complete and overall response rate to gemcitabine and docetaxel versus gemcitabine and irinotecan in chemotherapy naive patients with stage IIIB or IV non-small cell lung cancer. II. Compare the overall and failure free survival, duration of response, and toxicity associated with these combination regimens in this patient population.

OUTLINE: This is a randomized study. Patients are stratified according to disease stage (stage IIIB vs stage IV without CNS involvement vs stage IV with CNS involvement vs recurrent/progressive disease post surgery and/or radiotherapy). Patients are randomized to one of two treatment arms. Arm I: Patients receive gemcitabine IV over 30 minutes immediately followed by irinotecan IV over 90 minutes on days 1 and 8. Arm II: Patients receive gemcitabine IV over 30 minutes immediately followed by docetaxel IV over 60 minutes on days 1 and 8. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients achieving partial or complete response or stable disease receive treatment for least 6 courses and for 2 additional courses beyond the maximum response, and then at the investigator's discretion. Patients are followed every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter until disease progression or death.

PROJECTED ACCRUAL: A total of 72 patients (36 per treatment arm) will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed stage IIIB, IV, or recurrent non-small cell lung cancer (NSCLC) including: Squamous cell carcinoma Adenocarcinoma (including bronchoalveolar cell) Large cell anaplastic carcinoma (including giant and clear cell carcinomas) Stage IIIB eligible for other CALGB protocols consisting of combined chemotherapy and chest radiotherapy not permitted Malignant pleural effusion allowed CNS metastases allowed following completion of cranial radiotherapy Unidimensionally or bidimensionally measurable disease Solid tumor mass or hilar lesion surrounded by aerated lung Pleural based mass Mediastinal or hilar adenopathy clearly measurable No bone only disease No pleural or pericardial effusions No irradiated lesions unless progression is documented following radiotherapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.5 mg/dL SGOT no greater than 2 times upper limit of normal (ULN) Alkaline phosphatase less than 2.5 times ULN if SGOT is greater than 1.5 times ULN Renal: Creatinine no greater than 2.0 mg/dL Other: No other malignancies within the past 5 years except curatively treated basal or squamous cell skin cancer or carcinoma in situ of the cervix or breast Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics No prior chemotherapy for NSCLC Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics At least 2 weeks since prior radiotherapy At least 2 weeks since prior whole brain radiotherapy or stereotactic radiotherapy for CNS disease Surgery: At least 2 weeks since prior surgery for CNS disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 1999-09; Primary Completion 2004-07 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
response rate | Up to 2 years
overall survival | Up to 2 years
failure-free survival | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Caio Max S. Rocha Lima, MD, Study Chair — Medical University of South Carolina
Locations (8):
- United States (8):
  - Vincent T. Lombardi Cancer Research Center, Georgetown University, Washington D.C., District of Columbia
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Barnes-Jewish Hospital, St Louis, Missouri
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - University of Tennessee, Memphis Cancer Center, Memphis, Tennessee

REFERENCES:
- [Result] Rocha Lima CM, Rizvi NA, Zhang C, Herndon JE 2nd, Crawford J, Govindan R, King GW, Green MR; Cancer Leukemia Group B. Randomized phase II trial of gemcitabine plus irinotecan or docetaxel in stage IIIB or stage IV NSCLC. Ann Oncol. 2004 Mar;15(3):410-8. doi: 10.1093/annonc/mdh104. PMID 14998842
- [Result] Rocha Lima CM, Rizvi NA, Zhang K, et al.: CALGB 39809: Randomized phase II trial of gemcitabine/irinotecan and gemcitabine/docetaxel in stage IIIB (malignant pleural effusion) or stage IV NSCLC. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-1344, 2002.